CLINICAL TRIAL: NCT07358858
Title: A Randomized, Open-label, Two-period, Crossover Food Effect Study of QLS1410 in Healthy Chinese Adults
Brief Title: A Food Effect Study of QLS1410 in Healthy Chinese Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QSL1410-102
Record Dates: First submitted 2026-01-07; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Uncontrolled Hypertension

STUDY DESIGN:
Intervention Model Description: Model Description
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS1410 20mg (Experimental)
  Interventions: Drug: QLS1410

INTERVENTIONS:
Drug: QLS1410 — QLS1410 tablets

SUMMARY:
This study is aimed to evaluate the effect of food on pharmacokinetics of QLS1410 in healthy Chinese adults.

DETAILED DESCRIPTION:
All the qualified participants will be randomized (1:1) to two treatment sequences (fed/fasting and fasting/fed). In each period, participants will receive a single dosing of QLS1410 tablets either with or without a high-fat breakfast. There will be a one-week washout period in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to comply with all study visits, procedures, restrictions and provide the written informed consent form (ICF).
2. Males and females aged 18 to 55 years, inclusive.
3. Weight ≥ 50 kg for males and ≥ 45 kg for females, Body mass index (BMI) between 18 and 26 kg/m^2, inclusive, at screening.
4. Has a mean seated office systolic blood pressure (SBP) 110~139 mmHg (inclusive) and diastolic blood pressure (DBP) 70~89 mmHg (inclusive) at screening and baseline; measured 3 times consecutively (1-2 min intervals).
5. QTcF (QT corrected using Fridericia's formula) <450 ms for males and <470 ms for females.
6. Participants (including partners) must agree to abstain from sperm/egg donation and pregnancy plans, and to use highly effective contraception, from signing the ICF until 3 months after receiving the last dose of investigational product.

Exclusion Criteria:

1. Any medical condition/disease at screening deemed by the investigator to require exclusion, including but not limited to the cardiovascular, respiratory, digestive, urinary, endocrine metabolic, skeletal, muscular, hematologic, immune, nervous system.
2. Dysphagia or any surgical condition/disease that may affect drug absorption, distribution, metabolism, or excretion, at screening.
3. Use of systemic corticosteroids within 3 months prior to screening.
4. Any clinically significant abnormal result of vital signs, physical examinations, laboratory tests, chest X-ray, and abdominal B-ultrasound, at screening.
5. Active viral hepatitis (B or C), TP, and HIV as demonstrated by positive serology at Screening.
6. Mean pulse >100 or <50 bpm after ≥5 min of rest at screening (measured 3 times consecutively).
7. Any of the following laboratory abnormalities at screening: ALT or AST >1.5 x upper limit of normal (ULN); Total bilirubin >1.5 x ULN (participants with Gilbert's syndrome may qualify if direct bilirubin ≤ULN); Creatinine >ULN or eGFR <90 mL/min/1.73 m²; Serum potassium >ULN or sodium <135 mmol/L.
8. Smoking >5 cigarettes/day on average within 6 months before screening, or current use of e-cigarettes.
9. Alcohol consumption >14 units/week (1 unit = 357 mL of 3.5% beer, 27 mL of 40% spirits, or 104 mL of 12% wine) within 6 months before screening, or has a positive breath alcohol test at screening.
10. Blood donation >400 mL within 3 months or >200 mL within 4 weeks before screening, or plan to donate blood during the study.
11. Use of strong CYP3A4 or CYP1A2 inhibitors within 7 days or 5 half-lives (whichever is longer) before screening. Use of strong CYP3A4 inducer within 14 days or 5 half-lives (whichever is longer) before screening.
12. Use of any prescription drugs, OTC drugs, traditional medicines, and dietary supplements within 2 weeks or 5 half-lives (whichever is longer) prior to randomization.
13. Pregnant/lactating females or positive pregnancy test at screening.
14. Inability to tolerate a high-fat meal.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-23 (Estimated); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-02-07 (Estimated)

PRIMARY OUTCOMES:
AUC0-∞ | 0 to 96 hours
Area under the curve plasma concentration from time zero to Time of Last Quantifiable Concentration | 0 to 96 hours
Maximum observed plasma concentration | 0 to 96 hours